CLINICAL TRIAL: NCT01947582
Title: The Effects of Ankle Foot Orthoses (AFOs) on Mobility in Persons With Multiple Sclerosis (MS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Karen McCain, Associate Professor, School of Health Professions, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS Bracing
Record Dates: First submitted 2013-09-17; First posted 2013-09-20 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; gait; ankle foot orthosis (AFO)
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Application of ankle foot orthosis (Other): All participants will receive ankle foot orthosis or orthoses. Outcomes will be compared to pre-bracing findings.
  Interventions: Device: Ankle foot orthosis

INTERVENTIONS:
Device: Ankle foot orthosis — The ankle foot orthoses (AFOs) that will be used are designed to provide assistance with anterior tibial advancement during stance and dorsi flexion assistance during swing. The device(s) are polypropylene and are custom-fabricated.

SUMMARY:
The purpose of this study is to investigate the impact of ankle foot orthoses (AFOs) on the spatial and temporal gait parameters, electromyography (EMG), walking endurance, and quality of life in select individuals living with MS. The hypotheses of the study are: 1. Individuals who are fit with an AFO will demonstrate improvements in spatial and temporal gait parameters 2. Individuals who are fit with an AFO will demonstrate improvements in walking endurance. 3. Individuals who are fit with an AFO will demonstrate improvements in muscle firing profiles/EMG measures. 4. Individuals who are fit with an AFO will demonstrate improvements in quality of life.

DETAILED DESCRIPTION:
This is a non-randomized, single group (N=15), repeated measures study. The outcome measure for the study include: 1. GAITRite System for step length, 2. EMG of the anterior tibialis, gastrocnemius, soleus, and vastus lateralis muscles, 3. 6 Minute Walk Test (gait endurance) 4. 12-Item MS Walking Scale (Quality of Life assessment). This study will be 24 weeks long. Over the 24-week period, the subject will participate in 14 gait training sessions which will be at weeks 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 17, 20 and 23. The treatments will be 45-60 minutes in duration. Outcome measures (all or part) will be assessed at the following times: initial (T1), week 5 (T2), week 13 (T3), and week 24 (T4). Subjects will be closely monitored throughout the 24 week study and will be un-enrolled by self-request or the following medical reasons: 1. Acute exacerbation of MS symptoms, 2. New diagnosis with direct consequences affecting gait training, 3. Inability to tolerate the AFO.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a primary diagnosis of multiple sclerosis
* Individuals who are able to maintain a walking velocity of 30 cm/sec for at least 2 minutes independently or with the use of a single tip assistive device.
* Could have current or past history of single or bilateral AFO use, including neuroprostheses
* Evidence of weakness in plantarflexors

Exclusion Criteria:

* The presence of co-morbidities (neuromuscular or musculoskeletal) that would negatively impact gait training
* Individuals with BMI with >/= 40kg/m2
* Individuals with range of motion deficit in the ankle limiting passive range of motion to neutral dorsiflexion
* Individuals that plan to begin the use of Ampyra during the course of the study
* Individuals for whom the cost of an orthosis would represent a financial burden
* Individuals who are receiving concurrent physical therapy services elsewhere
* MSNQ of >22

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen J McCain, PT, DPT, NCS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center School of Health Professions, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Application of Ankle Foot Orthosis: persons in this group were fitted with bilateral ankle foot orthoses
Period: Overall Study
Arm/Group | Application of Ankle Foot Orthosis
Started | 2
Completed | 1
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Application of Ankle Foot Orthosis
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 48 [48 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Walking Distance During 6-Minute Walk Test
Description: Each participant walks at a self-selected velocity on level surfaces for 6 minutes. They will be allowed to use assistive devices if necessary. They will be asked to rate their level of exertion upon completion of walking on the rate of perceived exertion scale.
Time Frame: Assessed at visit 2 (week 1) and week 24
Measure: Number; unit: feet
Arm/Group | Application of Ankle Foot Orthosis
Number analyzed (Participants) | 1
feet | 222

2. Secondary Outcome: Change in Impact of MS on Fatigue Using the 12-Item Walk Scale
Description: The 12-Item Walk Scale is a paper and pencil test that asks persons with MS to rate their level of fatigue when doing functional tasks. The maximum possible score is 60 points and the lowest possible score is 12. Higher scores indicate a greater impact on walking than lower scores.
Time Frame: Assessed at visit 2 (week 1) and week 24
Measure: Number; unit: difference of sum of score
Arm/Group | Application of Ankle Foot Orthosis
Number analyzed (Participants) | 1
difference of sum of score | 1

3. Secondary Outcome: Change in Step Length Using the GAITRite Computerized Gait Analysis System
Description: Participants will be asked to walk on a 12-16 foot long vinyl pad placed on the floor.
Time Frame: Assessed at visit 2 (week 1) and week 24
Measure: Number; unit: cm
Arm/Group | Application of Ankle Foot Orthosis
Number analyzed (Participants) | 1
cm | 3.3

4. Secondary Outcome: Number of Persons With Change in Muscle Activity Using Surface Electromyography (EMG)
Description: Surface EMG is done on key muscles in the lower extremity (quadriceps, anterior tibialis, gastrocnemius, soleus) during computerized gait assessment. Changes in amplitude of muscle activity or timing of muscle activity would indicate, for example, increases in strength or changes in timing of muscles which might indicate motor learning as a result of wearing the ankle foot orthosis.
Time Frame: Assessed at visit 2 (week 1) and week 24
Measure: Number; unit: persons
Arm/Group | Application of Ankle Foot Orthosis
Number analyzed (Participants) | 1
persons | 1

ADVERSE EVENTS:
Arm/Group | Application of Ankle Foot Orthosis
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No